CLINICAL TRIAL: NCT03251248
Title: A Randomized, Double-blind, Crossover Study to Compare the Pharmacokinetic and Pharmacodynamic Bioequivalence of a Single Injection of MSB11455 and Neulasta in Healthy Adult Subjects
Brief Title: Pharmacokinetic/Pharmacodynamic Equivalence of MSB11455 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fresenius Kabi SwissBioSim GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: EMR200621-001
Record Dates: First submitted 2017-08-14; First posted 2017-08-16 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-01

CONDITIONS: Healthy
Keywords: MSB11455; Healthy subjects
MeSH Terms: interventions — pegfilgrastim

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- First MSB11455 Then Neulasta (Experimental)
  Interventions: Drug: MSB11455; Drug: Neulasta
- First Neulasta Then MSB11455 (Experimental)
  Interventions: Drug: MSB11455; Drug: Neulasta

INTERVENTIONS:
Drug: MSB11455 — Subjects will receive MSB11455 either on Period 1 Day 1 or Period 2 Day 1.
Drug: Neulasta — Subjects will receive Neulasta either on Period 1 Day 1 or Period 2 Day 1.
  Other Names: pegfilgrastim

SUMMARY:
The purpose of the study is to compare the pharmacokinetics (PK) and pharmacodynamics (PD) of MSB11455 and Neulasta in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who provide signed and dated written informed consent
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Subjects who have no known hypersensitivity to any component of Neulasta or MSB11455, and laboratory test results within predefined ranges
* Other protocol defined exclusion criteria could apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 294 (Actual)
Dates: Start 2017-08-22 (Actual); Primary Completion 2018-05-08 (Actual); Study Completion 2018-10-17 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve From Time Zero (Pre-dose) to Time of Last Quantifiable Concentration AUC(0-last) of MSB11455 and Neulasta | Pre-dose up to 15 days post-dose
Area Under the Concentration-Time Curve From Time Zero (Pre-dose) Extrapolated to Infinity AUC(0-inf) of MSB11455 and Neulasta | Pre-dose up to 15 days post-dose
Maximum Observed Plasma Concentration (Cmax) of MSB11455 and Neulasta | Pre-dose up to 15 days post-dose
Maximum Observed Effect (Emax) for Absolute Neutrophil Count (ANC) of MSB11455 and Neulasta | Pre-dose up to 15 days post-dose
Area Under the Effect-Time Curve From Time Zero (Pre-dose) to Last Measured Time (AUE0-t) for (ANC) of MSB11455 and Neulasta | Pre-dose up to 15 days post-dose

SECONDARY OUTCOMES:
Time to Maximum Observed Plasma Concentration (tmax) of MSB11455 and Neulasta | Pre-dose up to 15 days post-dose
Time to Last Observed Plasma Concentration (tlast) of MSB11455 and Neulasta | Pre-dose up to 15 days post-dose
Terminal rate constant (λz) of MSB11455 and Neulasta | Pre-dose up to 15 days post-dose
Terminal Half-life (t1/2) of MSB11455 and Neulasta | Pre-dose up to 15 days post-dose
Apparent Total Plasma Clearance (CL/F) of MSB11455 and Neulasta | Pre-dose up to 15 days post-dose
Time to Maximum Observed Effect (tEmax) for ANC of MSB11455 and Neulasta | Pre-dose up to 15 days post-dose
Area Under Effect Curve from zero to 360 hours (AUEC0-360) for ANC of MSB11455 and Neulasta | Pre-dose up to 15 days post-dose
Safety Profile as Assessed by Clinical Adverse events (AEs), Laboratory Variables, Vital Signs, Incidence of Antidrug Antibodies (ADAs), Neutralizing Antibodies(NABs) | Day 1 up to a maximum of 15 months
  Safety assessment will be based on number of subjects with AEs, abnormal laboratory variables, abnormal vital signs, incidence of ADAs and NABs

CONTACTS AND LOCATIONS:
Overall Officials: Radmila Kanceva, MD, PhD, Study Director — Fresenius Kabi SwissBioSim GmbH
Locations (2):
- Australia (2):
  - Nucleus Network, Melbourne, Victoria
  - Q-Pharm Pty Ltd, Herston

REFERENCES:
- [Derived] Lickliter J, Kanceva R, Vincent E, Schueler A, Harrison-Moench E, Yue CS, Stahl M, Ullmann M, Ghori V, Griffin P. Pharmacokinetics and Pharmacodynamics of a Proposed Pegfilgrastim Biosimilar MSB11455 Versus the Reference Pegfilgrastim Neulasta in Healthy Subjects: A Randomized, Double-blind Trial. Clin Ther. 2020 Aug;42(8):1508-1518.e1. doi: 10.1016/j.clinthera.2020.05.020. Epub 2020 Jul 11. PMID 32660769